CLINICAL TRIAL: NCT05255900
Title: Metabolic, Pressor and Neuropsychological Effects of Metyrapone Treatment in Patients With Hypercortisolism
Brief Title: Effects of Metyrapone in Patients With Hypercortisolism
Acronym: CEM
Status: Active, not recruiting | Type: Observational
Sponsor: Istituto Auxologico Italiano (Other)
Collaborators: HRA Pharma (Industry)
Responsible Party: Sponsor
Other Study IDs: 05J102
Record Dates: First submitted 2022-02-14; First posted 2022-02-25 (Actual); Last update posted 2025-09-08 (Actual); Status verified 2025-09

CONDITIONS: Hypercortisolism
Keywords: cortisol; metyrapone; hypercortisolism; mild hypercortisolism
MeSH Terms: conditions — Cushing Syndrome | interventions — Metyrapone

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- metyrapone treatment: hypercortisolemic patients taking metyrapone since less than a week (usually 250 mg/day, maximum dose 6000 mg/day)
  Interventions: Drug: Metyrapone Capsules

INTERVENTIONS:
Drug: Metyrapone Capsules — Exposure to 24 weeks of treatment with metyrapone

SUMMARY:
The aims of the present study are to evaluate in patients with mild hypercortisolism the effect of metyrapone treatment on glycometabolic control, blood pressure, thrombotic risk parameters, lipid profile, bone turnover markers, mental health and cortisol circadian rhythm.

DETAILED DESCRIPTION:
This open prospective observational study will include patients with mild hypercortisolism of both adrenal and pituitary origin not candidate for surgery. Patients taking metyrapone since less than a week will be followed up for 24 weeks. During this period of time, patients will be re-evaluated as far as blood pressure control, glycometabolic control, thrombotic risk parameters, lipid profile, bone turnover markers and cortisol circadian rhythm is concerned.

ELIGIBILITY:
Inclusion Criteria:

* Patients with mild Cushing's Syndrome not candidate for surgery
* Current therapy with metyrapone since less than 1 week
* Cortisol levels at 08:00 after 1 mg-overnight dexamethasone suppression test (1mgDST) >1.8 μg/dL
* Confirmed with 2 mg two days dexamethasone suppression test (2mgx2dDST)
* Presence of at least one out of the following conditions: type 2 diabetes mellitus, impaired fasting glucose (IFG) and/or impaired glucose tolerance (IGT), arterial hypertension, bone mineral density (BMD) Z-score < -2.0 and/or fragility fracture at any skeletal site
* Stable anti-hypertensive therapies and blood pressure (BP) levels in the month before enrolment
* Stable anti-diabetic therapies and glycometabolic control during the month before enrolment
* Stable body weight during the month before enrolment

Exclusion Criteria:

* Signs and/or symptoms of overt hypercortisolism (striae rubrae, moon facies, easy bruising, buffalo hump, hypertrichosis)
* Malignant hypertension and/or BP <200/120 mmHg
* Severe hyperglycemia (i.e. FG >350 mg/dL)
* Urinary free cortisol (UFC) higher than 1.5 fold the upper normal range
* Presence of pheochromocytoma or primary hyperaldosteronism
* Possible adrenal metastases or radiological features suggestive for adrenal malignancy (i.e. not homogeneous pattern, necrosis, calcifications, irregular margins, local invasion and high density at computed tomography)
* Congenital adrenal hyperplasia
* Intake of drugs influencing cortisol metabolism and/or secretion
* Women in child-bearing age
* Patients with body mass index (BMI) >35 kg/m2

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with hypercortisolism referred to the outpatient clinic who were already on metirapone therapy.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2022-04-28 (Actual); Primary Completion 2025-06-30 (Actual); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Proportion of patients with a mean systolic BP reduction of ≥5 mm Hg | Baseline, 24 weeks
  BP levels will be measured with arterial blood pressure monitoring (ABPM)

SECONDARY OUTCOMES:
Changes in glycometabolic control | 12 and 24 weeks
  i) the proportion of patients without type 2 diabetes achieving normalization of FG (<100 mg/dL) and/or the reduction of 2-hour glucose levels below 140 mg/dL after OGTT; ii) the proportion of patients with type 2 diabetes achieving HbA1c <7% among those with baseline HbA1c ≥7%;
Normalization of cortisol circadian rhythm | baseline, 12 weeks, 24 weeks.
  The cortisol circadian rhythm will be assessed by salivary cortisol levels determination (at 8 AM, 12 AM, 4 PM, 8 PM and 11 PM).
Changes of thrombotic risk parameters | Baseline, 12 and 24 weeks
  The thrombotic risk profile will be evaluated by measuring C-Protein, S-Protein, coagulation factor VIII and anti-thrombin III levels
Changes of lipid profile | Baseline, 12 and 24 weeks
  The lipid profile modifications will be evaluated by measuring total cholesterol, low-density lipoprotein, high-density lipoprotein and triglycerides
Changes of bone turnover markers | Baseline, 12 and 24 weeks
  The bone turnover changes will be assessed by measuring calcium, phosphorous, osteocalcin (OC), carboxy-terminal cross-linked telopeptide of type I collagen (CTX) and 24-h urinary calcium/creatinine ratio
Amelioration of psychological symptoms | Baseline, 12 and 24 weeks
  Psychological symptoms wil be evaluated with Beck Depression Inventory-II (BDI-II), a 21-item self-administered inventory designed to measure the intensity of depressive symptoms (Beck, Steer, & Brown, 1996). Scores ranging between 0 and 13 are indicative of minimal depression; scores that fall between 14 and 19 are considered to reflect a mild level of depression; scores of 20 to 28 are considered moderate; and a score ranging from 29 to 63 is labeled severe.

CONTACTS AND LOCATIONS:
Overall Officials: Chiodini Chiodini, Professor, Principal Investigator — Istituto Auxologico Italiano IRCCS
Locations (1):
- Istituto Auxologico Italiano, Milan, Italy

REFERENCES:
- [Background] Zavatta G, Di Dalmazi G. Recent Advances on Subclinical Hypercortisolism. Endocrinol Metab Clin North Am. 2018 Jun;47(2):375-383. doi: 10.1016/j.ecl.2018.01.003. Epub 2018 Apr 9. PMID 29754638
- [Background] Chiodini I, Morelli V. Subclinical Hypercortisolism: How to Deal with It? Front Horm Res. 2016;46:28-38. doi: 10.1159/000443862. Epub 2016 May 17. PMID 27212038
- [Background] Chiodini I. Clinical review: Diagnosis and treatment of subclinical hypercortisolism. J Clin Endocrinol Metab. 2011 May;96(5):1223-36. doi: 10.1210/jc.2010-2722. Epub 2011 Mar 2. PMID 21367932
- [Background] Morelli V, Arosio M, Chiodini I. Cardiovascular mortality in patients with subclinical Cushing. Ann Endocrinol (Paris). 2018 Jun;79(3):149-152. doi: 10.1016/j.ando.2018.03.005. Epub 2018 Mar 30. PMID 29606280
- [Background] Patrova J, Kjellman M, Wahrenberg H, Falhammar H. Increased mortality in patients with adrenal incidentalomas and autonomous cortisol secretion: a 13-year retrospective study from one center. Endocrine. 2017 Nov;58(2):267-275. doi: 10.1007/s12020-017-1400-8. Epub 2017 Sep 8. PMID 28887710
- [Background] Di Dalmazi G, Vicennati V, Garelli S, Casadio E, Rinaldi E, Giampalma E, Mosconi C, Golfieri R, Paccapelo A, Pagotto U, Pasquali R. Cardiovascular events and mortality in patients with adrenal incidentalomas that are either non-secreting or associated with intermediate phenotype or subclinical Cushing's syndrome: a 15-year retrospective study. Lancet Diabetes Endocrinol. 2014 May;2(5):396-405. doi: 10.1016/S2213-8587(13)70211-0. Epub 2014 Jan 29. PMID 24795253
- [Background] Debono M, Bradburn M, Bull M, Harrison B, Ross RJ, Newell-Price J. Cortisol as a marker for increased mortality in patients with incidental adrenocortical adenomas. J Clin Endocrinol Metab. 2014 Dec;99(12):4462-70. doi: 10.1210/jc.2014-3007. PMID 25238207
- [Background] Morelli V, Reimondo G, Giordano R, Della Casa S, Policola C, Palmieri S, Salcuni AS, Dolci A, Mendola M, Arosio M, Ambrosi B, Scillitani A, Ghigo E, Beck-Peccoz P, Terzolo M, Chiodini I. Long-term follow-up in adrenal incidentalomas: an Italian multicenter study. J Clin Endocrinol Metab. 2014 Mar;99(3):827-34. doi: 10.1210/jc.2013-3527. Epub 2014 Jan 1. PMID 24423350
- [Background] Park J, De Luca A, Dutton H, Malcolm JC, Doyle MA. Cardiovascular Outcomes in Autonomous Cortisol Secretion and Nonfunctioning Adrenal Adenoma: A Systematic Review. J Endocr Soc. 2019 Mar 25;3(5):996-1008. doi: 10.1210/js.2019-00090. eCollection 2019 May 1. PMID 31065617
- [Background] Chiodini I, Vainicher CE, Morelli V, Palmieri S, Cairoli E, Salcuni AS, Copetti M, Scillitani A. MECHANISMS IN ENDOCRINOLOGY: Endogenous subclinical hypercortisolism and bone: a clinical review. Eur J Endocrinol. 2016 Dec;175(6):R265-R282. doi: 10.1530/EJE-16-0289. Epub 2016 Jul 13. PMID 27412441
- [Background] Morelli V, Ghielmetti A, Caldiroli A, Grassi S, Siri FM, Caletti E, Mucci F, Aresta C, Passeri E, Pugliese F, Di Giorgio A, Corbetta S, Scillitani A, Arosio M, Buoli M, Chiodini I. Mental Health in Patients With Adrenal Incidentalomas: Is There a Relation With Different Degrees of Cortisol Secretion? J Clin Endocrinol Metab. 2021 Jan 1;106(1):e130-e139. doi: 10.1210/clinem/dgaa695. PMID 33017843
- [Background] Li D, Kaur RJ, Zhang CD, Ebbehoj A, Singh S, Atkinson EJ, Achenbach SJ, Rocca W, Khosla S, Bancos I. Risk of bone fractures after the diagnosis of adrenal adenomas: a population-based cohort study. Eur J Endocrinol. 2021 Apr;184(4):597-606. doi: 10.1530/EJE-20-1396. PMID 33606665
- [Background] Terzolo M, Pia A, Reimondo G. Subclinical Cushing's syndrome: definition and management. Clin Endocrinol (Oxf). 2012 Jan;76(1):12-8. doi: 10.1111/j.1365-2265.2011.04253.x. PMID 21988204
- [Background] Vassiliadi DA, Partsalaki E, Tsagarakis S. Approach to patients with bilateral adrenal incidentalomas. Curr Opin Endocrinol Diabetes Obes. 2020 Jun;27(3):125-131. doi: 10.1097/MED.0000000000000536. PMID 32209820
- [Background] Vassiliadi DA, Ntali G, Vicha E, Tsagarakis S. High prevalence of subclinical hypercortisolism in patients with bilateral adrenal incidentalomas: a challenge to management. Clin Endocrinol (Oxf). 2011 Apr;74(4):438-44. doi: 10.1111/j.1365-2265.2010.03963.x. PMID 21175735
- [Background] Vassilatou E, Vryonidou A, Ioannidis D, Paschou SA, Panagou M, Tzavara I. Bilateral adrenal incidentalomas differ from unilateral adrenal incidentalomas in subclinical cortisol hypersecretion but not in potential clinical implications. Eur J Endocrinol. 2014 Jul;171(1):37-45. doi: 10.1530/EJE-13-0848. Epub 2014 Apr 17. PMID 24743396
- [Background] Pasternak JD, Seib CD, Seiser N, Tyrell JB, Liu C, Cisco RM, Gosnell JE, Shen WT, Suh I, Duh QY. Differences Between Bilateral Adrenal Incidentalomas and Unilateral Lesions. JAMA Surg. 2015 Oct;150(10):974-8. doi: 10.1001/jamasurg.2015.1683. PMID 26200882
- [Background] Morelli V, Palmieri S, Salcuni AS, Eller-Vainicher C, Cairoli E, Zhukouskaya V, Scillitani A, Beck-Peccoz P, Chiodini I. Bilateral and unilateral adrenal incidentalomas: biochemical and clinical characteristics. Eur J Endocrinol. 2013 Jan 17;168(2):235-41. doi: 10.1530/EJE-12-0777. Print 2013 Feb. PMID 23169694
- [Background] Toini A, Dolci A, Ferrante E, Verrua E, Malchiodi E, Sala E, Lania AG, Chiodini I, Beck-Peccoz P, Arosio M, Spada A, Mantovani G. Screening for ACTH-dependent hypercortisolism in patients affected with pituitary incidentaloma. Eur J Endocrinol. 2015 Apr;172(4):363-9. doi: 10.1530/EJE-14-0599. PMID 25722096
- [Background] Chiodini I, Albani A, Ambrogio AG, Campo M, De Martino MC, Marcelli G, Morelli V, Zampetti B, Colao A, Pivonello R; ABC Group. Six controversial issues on subclinical Cushing's syndrome. Endocrine. 2017 May;56(2):262-266. doi: 10.1007/s12020-016-1017-3. Epub 2016 Jul 12. PMID 27406391
- [Background] Fassnacht M, Dekkers OM, Else T, Baudin E, Berruti A, de Krijger R, Haak HR, Mihai R, Assie G, Terzolo M. European Society of Endocrinology Clinical Practice Guidelines on the management of adrenocortical carcinoma in adults, in collaboration with the European Network for the Study of Adrenal Tumors. Eur J Endocrinol. 2018 Oct 1;179(4):G1-G46. doi: 10.1530/EJE-18-0608. PMID 30299884
- [Background] Bancos I, Alahdab F, Crowley RK, Chortis V, Delivanis DA, Erickson D, Natt N, Terzolo M, Arlt W, Young WF Jr, Murad MH. THERAPY OF ENDOCRINE DISEASE: Improvement of cardiovascular risk factors after adrenalectomy in patients with adrenal tumors and subclinical Cushing's syndrome: a systematic review and meta-analysis. Eur J Endocrinol. 2016 Dec;175(6):R283-R295. doi: 10.1530/EJE-16-0465. Epub 2016 Jul 22. PMID 27450696
- [Background] Salcuni AS, Morelli V, Eller Vainicher C, Palmieri S, Cairoli E, Spada A, Scillitani A, Chiodini I. Adrenalectomy reduces the risk of vertebral fractures in patients with monolateral adrenal incidentalomas and subclinical hypercortisolism. Eur J Endocrinol. 2016 Mar;174(3):261-9. doi: 10.1530/EJE-15-0977. Epub 2015 Dec 2. PMID 26630908
- [Background] Papierska L, Cwikla J, Rabijewski M, Glinicki P, Otto M, Kasperlik-Zaluska A. Adrenal (131)I-6beta-iodomethylnorcholesterol scintigraphy in choosing the side for adrenalectomy in bilateral adrenal tumors with subclinical hypercortisolemia. Abdom Imaging. 2015 Oct;40(7):2453-60. doi: 10.1007/s00261-015-0452-6. PMID 26041277
- [Background] Albiger NM, Ceccato F, Zilio M, Barbot M, Occhi G, Rizzati S, Fassina A, Mantero F, Boscaro M, Iacobone M, Scaroni C. An analysis of different therapeutic options in patients with Cushing's syndrome due to bilateral macronodular adrenal hyperplasia: a single-centre experience. Clin Endocrinol (Oxf). 2015 Jun;82(6):808-15. doi: 10.1111/cen.12763. Epub 2015 Mar 27. PMID 25727927
- [Background] Donadio F, Morelli V, Salcuni AS, Eller-Vainicher C, Carletto M, Castellani M, Dellavedova L, Scillitani A, Beck-Peccoz P, Chiodini I. Role of adrenal gland scintigraphy in patients with subclinical hypercortisolism and incidentally discovered adrenal mass. J Endocrinol Invest. 2009 Jul;32(7):576-80. doi: 10.1007/BF03346511. Epub 2009 Jun 15. PMID 19535891
- [Background] Debillon E, Velayoudom-Cephise FL, Salenave S, Caron P, Chaffanjon P, Wagner T, Massoutier M, Lambert B, Benoit M, Young J, Tabarin A, Chabre O. Unilateral Adrenalectomy as a First-Line Treatment of Cushing's Syndrome in Patients With Primary Bilateral Macronodular Adrenal Hyperplasia. J Clin Endocrinol Metab. 2015 Dec;100(12):4417-24. doi: 10.1210/jc.2015-2662. Epub 2015 Oct 9. PMID 26451908
- [Background] Giovanelli L, Aresta C, Favero V, Bonomi M, Cangiano B, Eller-Vainicher C, Grassi G, Morelli V, Pugliese F, Falchetti A, Gennari L, Scillitani A, Persani L, Chiodini I. Hidden hypercortisolism: a too frequently neglected clinical condition. J Endocrinol Invest. 2021 Aug;44(8):1581-1596. doi: 10.1007/s40618-020-01484-2. Epub 2021 Jan 4. PMID 33394454
- [Background] Feelders RA, Newell-Price J, Pivonello R, Nieman LK, Hofland LJ, Lacroix A. Advances in the medical treatment of Cushing's syndrome. Lancet Diabetes Endocrinol. 2019 Apr;7(4):300-312. doi: 10.1016/S2213-8587(18)30155-4. Epub 2018 Jul 20. PMID 30033041
- [Background] Puglisi S, Perotti P, Barbot M, Cosio P, Scaroni C, Stigliano A, Lardo P, Morelli V, Polledri E, Chiodini I, Reimondo G, Pia A, Terzolo M. Preoperative treatment with metyrapone in patients with Cushing's syndrome due to adrenal adenoma: a pilot prospective study. Endocr Connect. 2018 Nov;7(11):1227-1235. doi: 10.1530/EC-18-0400. PMID 30352400
- [Background] Daniel E, Newell-Price JD. Therapy of endocrine disease: steroidogenesis enzyme inhibitors in Cushing's syndrome. Eur J Endocrinol. 2015 Jun;172(6):R263-80. doi: 10.1530/EJE-14-1014. Epub 2015 Jan 30. PMID 25637072
- [Background] Daniel E, Aylwin S, Mustafa O, Ball S, Munir A, Boelaert K, Chortis V, Cuthbertson DJ, Daousi C, Rajeev SP, Davis J, Cheer K, Drake W, Gunganah K, Grossman A, Gurnell M, Powlson AS, Karavitaki N, Huguet I, Kearney T, Mohit K, Meeran K, Hill N, Rees A, Lansdown AJ, Trainer PJ, Minder AE, Newell-Price J. Effectiveness of Metyrapone in Treating Cushing's Syndrome: A Retrospective Multicenter Study in 195 Patients. J Clin Endocrinol Metab. 2015 Nov;100(11):4146-54. doi: 10.1210/jc.2015-2616. Epub 2015 Sep 9. PMID 26353009
- [Background] Debono M, Harrison RF, Chadarevian R, Gueroult C, Abitbol JL, Newell-Price J. Resetting the Abnormal Circadian Cortisol Rhythm in Adrenal Incidentaloma Patients With Mild Autonomous Cortisol Secretion. J Clin Endocrinol Metab. 2017 Sep 1;102(9):3461-3469. doi: 10.1210/jc.2017-00823. PMID 28911138
- [Background] Lombardo G, Enache D, Gianotti L, Schatzberg AF, Young AH, Pariante CM, Mondelli V. Baseline cortisol and the efficacy of antiglucocorticoid treatment in mood disorders: A meta-analysis. Psychoneuroendocrinology. 2019 Dec;110:104420. doi: 10.1016/j.psyneuen.2019.104420. Epub 2019 Aug 23. PMID 31499391
- [Background] Sigalas PD, Garg H, Watson S, McAllister-Williams RH, Ferrier IN. Metyrapone in treatment-resistant depression. Ther Adv Psychopharmacol. 2012 Aug;2(4):139-49. doi: 10.1177/2045125312436597. PMID 23983967
- [Background] Athimulam S, Delivanis D, Thomas M, Young WF, Khosla S, Drake MT, Bancos I. The Impact of Mild Autonomous Cortisol Secretion on Bone Turnover Markers. J Clin Endocrinol Metab. 2020 May 1;105(5):1469-77. doi: 10.1210/clinem/dgaa120. PMID 32154561
- [Background] Unger T, Borghi C, Charchar F, Khan NA, Poulter NR, Prabhakaran D, Ramirez A, Schlaich M, Stergiou GS, Tomaszewski M, Wainford RD, Williams B, Schutte AE. 2020 International Society of Hypertension Global Hypertension Practice Guidelines. Hypertension. 2020 Jun;75(6):1334-1357. doi: 10.1161/HYPERTENSIONAHA.120.15026. Epub 2020 May 6. No abstract available. PMID 32370572
- [Background] Inzucchi SE, Bergenstal RM, Buse JB, Diamant M, Ferrannini E, Nauck M, Peters AL, Tsapas A, Wender R, Matthews DR; American Diabetes Association (ADA); European Association for the Study of Diabetes (EASD). Management of hyperglycemia in type 2 diabetes: a patient-centered approach: position statement of the American Diabetes Association (ADA) and the European Association for the Study of Diabetes (EASD). Diabetes Care. 2012 Jun;35(6):1364-79. doi: 10.2337/dc12-0413. Epub 2012 Apr 19. No abstract available. PMID 22517736
- [Background] Singh B, Saxena A. Surrogate markers of insulin resistance: A review. World J Diabetes. 2010 May 15;1(2):36-47. doi: 10.4239/wjd.v1.i2.36. PMID 21537426